CLINICAL TRIAL: NCT04846127
Title: A Multi-Center Registry Evaluating Participants Who Receive CanGaroo® Envelope or No Envelope During CIED Implantation
Brief Title: CanGaroo® Registry Study
Status: Completed | Type: Observational
Sponsor: Elutia Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: CPR-2218
Record Dates: First submitted 2021-04-12; First posted 2021-04-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Arrhythmias, Cardiac
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- CanGaroo Envelope: Participants who receive a CanGaroo envelope during their CIED implant.
  Interventions: Device: CanGaroo Envelope
- No Envelope: Participants who do not receive an envelope of any kind during their CIED implant.

INTERVENTIONS:
Device: CanGaroo Envelope — Utilization of a CanGaroo envelope with the CIED during the participant's CIED implant procedure.
  Groups: CanGaroo Envelope

SUMMARY:
A Multi-Center Registry Evaluating Participants Who Receive CanGaroo Envelope or No Envelope During their CIED Implantation

DETAILED DESCRIPTION:
This prospective, multi-center study will enroll up to 500 participants who are undergoing their initial CIED implant with either a CanGaroo envelope or no envelope.

Once a participant is enrolled in one of the two cohorts, each participant will have their medical history data reviewed and data will be recorded in the CRF including baseline demographics, medications, and diagnoses.

The details of the CIED procedure including any complications/AEs that occur during the procedure will be captured on the appropriate CRF.

Information collected at the follow-up visits will include documentation of post-procedure status, including any complications, adverse events, or revision/reoperation procedures that occur during the follow-up period. This information will also be collected for any unscheduled follow-ups, visits, or care encounters that occur up to 3 months post-procedure. For participants that agree and qualify for optional long-term follow-up, the same information will be collected at additional follow-up points every six months for up to five years.

ELIGIBILITY:
Inclusion Criteria:

1. Participants for whom this is their first CIED implantation at a particular anatomical site.

   Participants with a history of prior CIED implants at other anatomical sites than the current site can be included, provided that the planned implant location for the current CIED procedure is the first implant procedure at that site.
2. Participants aged 18 years or older at time of enrollment.
3. Participant is able and agrees to provide written informed consent and use of PHI.

Exclusion Criteria:

1. Participants who have had one or more prior CIED procedures (implantations or revisions) at the current device implant site.
2. Participants under the age of 18 at time of enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 500 participants who will either receive a CanGaroo envelope or no envelope during their de novo cardiac implantable electronic device implantation.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2023-04-17 (Actual); Study Completion 2024-10-17 (Actual)

PRIMARY OUTCOMES:
Association between participant characteristics and outcomes | 3 months post-procedure
  Cohort comparison of clinically significant factors such as physical and demographic characteristics, medical history risk factors related to post-procedure events, and associations with outcomes and events.
Association between CanGaroo envelope use and CIED implant-related outcomes and events. | 3 months post-procedure
  Cohort comparison of clinically significant events such as infection, wound healing issues, CIED migration, CIED erosion, or a revision/reoperation procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas F. Deering, MD, Principal Investigator — Piedmont Heart Institute
Locations (23):
- United States (23):
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Daytona Heart Group, Daytona Beach, Florida
  - The Arrhythmia Center of South Florida, Delray Beach, Florida
  - Florida Heart Rhythm Specialists, PLLC, Fort Lauderdale, Florida
  - VA Medical Center, Gainesville, Florida
  - Cardiovascular Associates/Osceola Regional Medical Center, Kissimmee, Florida
  - Advent Health, Tampa, Florida
  - Baptist Health Floyd, New Albany, Indiana
  - St. Joseph Hospital, Lexington, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Brigham & Women's Hospital, Cardiovascular Division, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Ascension Providence Hospital, Southfield, Michigan
  - Metro Health/University of Michigan Health, Wyoming, Michigan
  - UNC Health/NC Heart & Vascular Research, Raleigh, North Carolina
  - New Hanover Regional Medical Center, Wilmington, North Carolina
  - Mercy Health, Toledo, Ohio
  - Oklahoma State University Center for Health Sciences, Tulsa, Oklahoma
  - University of Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Carolina Heart Specialists, Lancaster, South Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - Houston Methodist, Houston, Texas
  - Heart Rhythm Associates, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Aziyo Biologics, Inc. website — http://aziyo.com